CLINICAL TRIAL: NCT00140790
Title: Effects of Valsartan on Cardiovascular Events in Patients With Renal Dysfunction
Brief Title: Valsartan in Cardiovascular Disease With Renal Dysfunction (The V-CARD) Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The number of actual events was extremely low. We extended the study period, but it was still not enough. Also, many patients were loss of follow up.
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Hisao Ogawa, Professor, Kumamoto University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CVM-RCT-2005-02
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Hypertension
Keywords: Cardiorenal syndrome; Renal dysfunction; Cardiovascular events; Valsartan
MeSH Terms: conditions — Hypertension; Cardio-Renal Syndrome; Renal Insufficiency | interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valsartan 40mg (Active Comparator): Standard Dose valsartan
  Interventions: Drug: valsartan
- Valsartan 160mg (Active Comparator): High Dose valsartan
  Interventions: Drug: valsartan

INTERVENTIONS:
Drug: valsartan — valsartan 40 or 160 (80) mg per day

SUMMARY:
The purpose of this study is to investigate if an angiotensin II receptor blocker, valsartan 160 mg/day is more effective to reduce the incidence of cardiovascular events as compared to 40 mg/day in patients with moderate renal dysfunction.

DETAILED DESCRIPTION:
It is well known that patients with renal dysfunction have a poor prognosis concerning cardiovascular diseases. That is called "cardiorenal syndrome". It was reported that valsartan was effective in reducing the urine albumin extraction rate in patients with hyper- or normotension. We hypothesized that valsartan was more effective to prevent cardiovascular events by the intermediary of improving renal function.

The primary endpoints are:

* cardiovascular events (cardiac death, non-fatal myocardial infarction, unstable angina requiring rehospitalization, congestive heart failure requiring rehospitalization, revascularization procedures including coronary angioplasty or coronary artery bypass grafting;Stroke or transient ischaemic attack, dissociation aneurysm of the aorta needing hospitalisation;Lower limbs artery obstruction needing hospitalisation .
* end-stage renal dysfunction (introduction of hemodialysis or kidney transplantation)
* 50% reduction of creatinine clearance

The secondary endpoints are:

* systolic and diastolic function of the left ventricle estimated by echocardiography (% FS and E/A ratio)
* specific biochemical markers for cardiac or renal function (urine microalbumin, plasma B-type natriuretic peptide, plasma type 1 plasminogen activator inhibitor, plasma cystatin C)
* % changes of creatinine clearance between start and end of the study period
* transition of 1/(serum Cr) in patients whose u-prot/u-Cr is equal to or more than 1.0
* transition of serum K
* HbA1c
* New onset Atrial Fibrillation
* New onset Diabetes

ELIGIBILITY:
Inclusion Criteria (all required):

* Systolic blood pressure (SBP) >/= 140 and/or diastolic blood pressure (DBP) >/= 90 (untreated hypertension cases); or SBP>/=130 and/or DBP>/=80 (treated hypertension cases)
* Patients with coronary artery disease (more than 50% stenosis on coronary angiography [CAG], coronary computed tomography [CT] or coronary magnetic resonance angiography [MRA]; coronary spasm; or history of percutaneous coronary intervention [PCI]);Unstable angina patient
* Creatinine clearance between 30.0 and 89.9 ml/min

Exclusion Criteria (at least one of following):

* Reduced left ventricular (LV) function (ejection fraction [EF] equal to or less than 40%)
* Hyperpotassemia (serum potassium equal to or more than 5.5 mEq/l)
* Rapid progressive glomerular nephritis
* Nephrotic syndrome
* Renal artery stenosis
* Uncontrolled diabetes (HbA1c equal to or more than 9.0%)
* History of allergy to valsartan
* Pregnant women

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2006-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Cardiovascular events | 2 years
End-stage renal dysfunction | 2 years
50% reduction of creatinine clearance | 2 years

SECONDARY OUTCOMES:
% FS and E/A ratio | 2 years
Specific biochemical markers for cardiac or renal function | 6 months and 1 year and 2 years
% changes of creatinine clearance | 2 years
1/(serum Cr) | 2 years
Serum K | 2 years
HbA1c | 2 years
U-prot/U-Cr | 2 years
Adverse drug effects | 2 years
New onset Atrial Fibrillation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hisao Ogawa, MD, PhD, Study Chair — Department of Cardiovascular Medicine, Graduate School of Medical Sciences, Kumamoto University
Locations (2):
- Japan (2):
  - Department of Cardiovascular Medicine, Kumamoto University Hospital, Kumamoto, Kumamoto
  - Department of Cardiovascular Medicine, Graduate School of Medical Sciences, Kumamoto University, Kumamoto